CLINICAL TRIAL: NCT00875719
Title: Comparing Effectiveness of Oxygen Supplementation From a Portable Concentrator and a Liquid Oxygen Source During Walking Test in COPD Patients With Respiratory Failure
Brief Title: Oxygen Portable Concentrator During Exercises in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche (Other)
Responsible Party: Jean François MUIR - President, ANTADIR
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANTADIR CMTS OXYGEN 2009
Record Dates: First submitted 2009-03-27; First posted 2009-04-03 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD patients with respiratory failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- continuous v intermittent Oxygen therapy (Active Comparator): intermittent oxygen compared to constant flow oxygen as regards walking distance
  Interventions: Device: Oxygen concentrators versus constant flow axygen; Device: oxygen concentrator

INTERVENTIONS:
Device: Oxygen concentrators versus constant flow axygen — Each patient performed 2 walking tests, and received oxygen supplementation from a portable concentrator or a liquid oxygen source, in a random order.
  Other Names: portable oxygen concentrator
Device: oxygen concentrator — comparison walk distance and saturation with continuous oxygen compared to intermittent oxygen
  Other Names: portable concentrator

SUMMARY:
The purpose of this study is to compare differences in oxygen delivery between portable oxygen concentrators (POCs) and liquid oxygen (LOs) portable units, pose a question if POCs are equally effective as LOs in reducing exercise-induced hypoxaemia. DESIGN: Randomized, single-blind clinical trial.

DETAILED DESCRIPTION:
Our primary objective is to compare at rest and during exercise the evolution of oxygen saturation and dyspnea during 6 minutes walking test in patients with COPD receiving oxygen supplementation either with portable concentrators or liquid oxygen in a random order.

ELIGIBILITY:
Inclusion Criteria:

* COPD with respiratory failure and indication for oxygen supplementation at rest and/or during exercice.

Exclusion Criteria:

* Evolutive heart disease.
* Unability to understand or realize the tests.
* Acute exacerbation during the last month.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Oxygen Saturation | One day

SECONDARY OUTCOMES:
Walking Distance | One day

CONTACTS AND LOCATIONS:
Overall Officials: Boris MELLONI, Pr, Principal Investigator — Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche
Locations (1):
- Service de Pneumologie et Allergologie- Hôpital le Cluzeau. 23 av. D. Larrey, Limoges, France